CLINICAL TRIAL: NCT03006120
Title: Treatment Management and Factors Affecting Mortality in Retroperitoneal Hemorrhage Due to Cardiac Catheterization; Single Center Experience
Status: Completed | Type: Observational
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ebubekir Gündeş, Director,Depertmant of Gastroenterological Surgery, Principal Investigator, Clinical M.D, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2016.5/7-18
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Treatment Procedure; Mortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Group 1: Conservative management
  Interventions: Procedure: Retroperitoneal hematoma due to cardiac catheterization
- Group 2: Angiografic stenting
  Interventions: Procedure: Retroperitoneal hematoma due to cardiac catheterization
- Group 3: Surgery
  Interventions: Procedure: Retroperitoneal hematoma due to cardiac catheterization

INTERVENTIONS:
Procedure: Retroperitoneal hematoma due to cardiac catheterization

SUMMARY:
Bleeding complications after cardiac catheterization have been reviewed previously, but there are very few studies on retroperitoneal hematoma and appropriate treatment of patients is not well defined. For this reason, the investigators aimed to analyze the clinical manifestations of retroperitoneal hematomas in a single center using a case-control study design, to analyze the treatment procedure determinants and consequently to provide an updated and usable treatment algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Retroperitoneal hematoma following cardiac catheterization

Exclusion Criteria:

* Patients with retroperitoneal hematomas other than cardiac catheterization and patients with missing file records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retroperitoneal hematoma following cardiac catheterization in our institution between January 2010 and October 2016.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 01/01/2010- 31/10/2016